

#### **Title Page** 1.0

# **Statistical Analysis Plan**

Study M16-004 (1311.38)

A Phase II/III, Randomized, Double-blind Study to **Evaluate Efficacy and Safety of Two Different Dose** Regimens of Risankizumab and Placebo and **Maintenance of Response of Risankizumab Administered Subcutaneously in Japanese Patients** With Moderate to Severe Chronic Plaque Type **Psoriasis** 

Date: 10 Jan 2018

Version 1.0

| 2.0 | Table of Contents | |
|---|---|---|
| 1.0 | Title Page | 1 |
| 2.0 | Table of Contents | 2 |
| 3.0 | Introduction | 5 |
| 4.0 | Study Objectives, Design and Procedures | 5 |
| 4.1 | Objectives | 5 |
| 4.2 | Design Diagram | 6 |
| 4.3 | Sample Size | 7 |
| 4.4 | Interim Analysis | 7 |
| 5.0 | Analysis Populations and Stratification | 8 |
| 5.1 | Analysis Populations | 8 |
| 5.2 | Variables Used for Stratification of Randomization | |
| 6.0 | Analysis Conventions | 10 |
| 7.0 | Demographics, Baseline Characteristics, Medical History, and Previous/Concomitant Medications | 16 |
| 7.1 | Demographic and Baseline Characteristics | 16 |
| 7.2 | Medical History | 18 |
| 7.3 | Previous Treatment and Concomitant Medications | 18 |
| 7.4 | Protocol Deviations | 19 |
| 8.0 | Patient Disposition | 19 |
| 9.0 | Study Drug Exposure and Compliance | 20 |
| 10.0 | Efficacy Analysis | 21 |
| 10.1 | General Considerations. | 21 |
| 10.1.1 | Analyses of Categorical Variables | 22 |
| 10.1.2 | Analyses of Continuous Variables | 23 |
| 10.1.3 | Analyses of Time-to-Event Variables | 24 |
| 10.1.4 | Missing Data Imputations | 25 |
| 10.1.5 | Analysis of Psoriasis Symptoms Scale (PSS) | 26 |
| 10.2 | Primary Efficacy Analysis | 27 |
| 10.3 | Secondary Efficacy Analyses | 28 |
| 10.3.1 | Further Efficacy Analysis | |
| 10.4 | Handling of Multiplicity | 30 |



Risankizumab
M16-004 – Statistical Analysis Plan
Version 1.0 – 10 Jan 2018

| 10.5 | Efficacy Subgroup Analysis | 31 |
|---|---|---|
| 11.0 | Safety Analysis | 31 |
| 11.1 | General Considerations. | 31 |
| 11.2 | Analysis of Adverse Events | 32 |
| 11.2.1 | Treatment-Emergent Adverse Events. | 32 |
| 11.2.2 | SAEs (Including Deaths) and Adverse Events Leading to Study<br>Drug Discontinuation | 40 |
| 11.2.3 | Safety Subgroup Analysis | 40 |
| 11.3 | Analysis of Laboratory Data | 41 |
| 11.3.1 | Variables and Criteria Defining Abnormality | 41 |
| 11.3.2 | Statistical Methods | 43 |
| 11.4 | Analysis of Vital Signs and Weight | 46 |
| 11.4.1 | Variables and Criteria Defining Abnormality | 46 |
| 11.4.2 | Statistical Methods | 47 |
| 11.5 | Analysis of ECG Parameters | 48 |
| 11.6 | Local Tolerability | 48 |
| 12.0 | Pharmacokinetic Analysis | 49 |
| 13.0 | Biomarkers Analysis | 49 |
| 14.0 | Summary of Changes | 49 |
| 14.1 | Summary of Changes Between the Latest Version of Protocol and the Current SAP | 49 |
| 14.2 | Summary of Changes Between the Previous Version and the Current Version of the SAP | 49 |
| 15.0 | Appendix | 49 |
| 16.0 | References | 49 |
| 17.0 | List of Tables, Figures, and Data Listings to Be<br>Programmed | 49 |
| List of Tabl | es | |
| Table 1. | Notation for Treatment Groups | 9 |
| Table 2. | Visit Windows for Analysis of PASI, Vital Signs, and Local Tolerability in Part A (ITT/PP/Safety Populations) | 13 |



Risankizumab M16-004 – Statistical Analysis Plan Version 1.0 – 10 Jan 2018

| Table 3. | Visit Windows for Analysis of Safety Laboratory Tests in Part A (Safety Population) | 13 |
|---|---|---|
| Table 4. | Visit Windows for Analysis of ECG in Part A (Safety Population) | 13 |
| Table 5. | Visit Windows for Analysis of sPGA, PSS, DLQI, HAQ-DI, Pain VAS, Investigator's Global Assessment VAS, Patient's Global Assessment VAS, CRP as an ACR 20 Component, SJC, and TJC in Part A (ITT Population) | 14 |
| Table 6. | Visit Windows for Analysis of PASI, Vital Signs, and Local Tolerability in Part B (ITT/Safety Population) | 14 |
| Table 7. | Visit Windows for Analysis of sPGA, PSS, DLQI, HAQ-DI, Pain VAS, Investigator's Global Assessment VAS, Patient's Global Assessment VAS, SJC, TJC, Laboratory Tests, and ECG in Part B (ITT/Safety Population) | 15 |
| Table 8. | Visit Windows for Summary of Study Drug Injections in Part A | 15 |
| Table 9. | Visit Windows for Summary of Study Drug Injections in Part B | 15 |
| Table 10. | Areas of Safety Interest | 36 |
| Table 11. | Clinical Laboratory Tests | 42 |
| Table 12. | Criteria for Potentially Clinically Important Chemistry Values | 44 |
| Table 13. | Criteria for Potentially Clinically Important Hematology Values | 44 |
| Table 14. | NCI CTCAE Grading | 45 |
| Table 15. | Criteria for Potentially Clinically Important Vital Sign Findings | 47 |
| List of Fig | gures | |
| Figure 1. | Study Design Schematic | 6 |



#### 3.0 Introduction

This Statistical Analysis Plan (SAP) describes the statistical analysis to be completed by the AbbVie Clinical Statistics Department for risankizumab study Protocol M16-004 (BI Study 1311.38) dated 05 September 2016 and the protocol amendment dated 07 June 2017.

This SAP will provide details to further elaborate statistical methods as outlined in the Protocol of Study 1311.38.

Analyses will be performed using SAS® version 9.4 (SAS. Institute, Inc., Cary, NC 27513) or higher using the UNIX operating system.

SAP will not be updated in case of future administrative or minor amendments to the protocol unless the changes have any impact on the analysis of the study data.

# 4.0 Study Objectives, Design and Procedures

# 4.1 Objectives

The objectives of this study are to assess the efficacy and safety of two different dose regimens of risankizumab compared to placebo in patients with moderate to severe chronic plaque psoriasis. The primary efficacy evaluation will be performed at Week 16 and an assessment of maintenance of response will be performed at Week 52.

In the subset of enrolled patients with concomitant psoriatic arthritis, the signs and symptoms of psoriatic arthritis will be evaluated to assess improvement during the trial.

This trial will assess PK and the emergence of anti-drug antibodies (ADA) and their effect on efficacy and safety. Moreover, it will be explored how the use of risankizumab may influence protein expression levels and disease specific protein markers. These analyses will not be covered in this SAP.

#### 4.2 Design Diagram

This randomized, double-blind, double-dummy, placebo controlled, parallel design study compares two different dose regiments of risankizumab with placebo. In total, approximately 168 patients with moderate to severe chronic plaque psoriasis will be randomized in this trial.

Patients are randomized at a ratio of 2:2:1:1 to one of 4 treatment arms (risankizumab 75 mg, risankizumab 150 mg, placebo switching to risankizumab 75 mg after Week 16, and placebo switching to risankizumab 150 mg after Week 16) as shown in Figure 1.

Randomization will be stratified by concomitant PsA at baseline (Yes versus No) and body weight ( $\leq$  90 kg versus > 90 kg).

Patients will be offered to roll over into an extension trial, if they have completed the study and meet the inclusion criteria for the extension trial.

N=56 BI 655066 (risankizumab) 75 mg (week 0, 4 then every 12 weeks) N=56 BI 655066 (risankizumab) 150 mg (week 0, 4 then every 12 weeks) R BI 655066 (risankizumab) 75 mg (every 12 weeks) Placebo (week 0, 4) N=28 Placebo (week 0, 4) N=28 BI 655066 (risankizumab) 150 mg (every 12 weeks) Wk16 Wk28 Wk40 Wk52 Wk4 WkO Wk56 =dosing visit at study Week (Wk) as labelled 1 =option to enter the extension trial

Figure 1. Study Design Schematic

BI 655066 is risankizumab.



#### 4.3 Sample Size

For the Japanese submission, the safety data of at least 100 Japanese patients exposed to risankizumab at the registered dose(s) for 1 year or more is necessary for long team safety assessment as a result of the PMDA consultation meeting in 2015. This study will enroll a total of 168 patients, with 56 patients in each of the two risankizumab arms and 56 patients in the placebo arm. It is expected that at least 68 patients exposed to risankizumab 75 mg and 68 patients exposed to risankizumab 150 mg will reach at least 1 year exposure to risankizumab in this clinical trial or in the following extension study. Other global phase 3 trials where Japanese patients are to be enrolled will make up for the remaining safety data requirements.

Based on the outcome from the Trial 1311.2, the PASI 90 response rate at Week 16 is assumed to be at least 65% in each of the risankizumab arm. The phase 3 results from ustekinumab and secukinumab indicate a response rate for PASI 90 of approximately 5% in the placebo arm. With hieratical order of testing the 150 mg risankizumab vs placebo followed 75 mg risankizumab vs placebo, the above sample size will provide more than 90% power to detect the superiority of both risankizumab arms vs placebo.

# 4.4 Interim Analysis

Before the submission to regulatory agencies with the long-term data, an interim report will be prepared for the submissions analysis pertaining to Part A. Primary endpoint (PASI 90 score at Week 16) for all patients will be included in the Week 28 analyses, which is the only and final analysis for the primary endpoint; hence no alpha adjustment is required. For this analysis all efficacy endpoints and safety as well as PK and immunogenicity data will be analysed. As endpoints for Week 28, same analyses will be performed for the Week 52 endpoints defined in Section 10.3.

AbbVie Data and Statistical Sciences will be unblinded to perform this analysis. Unblinded treatment assignments will not be disseminated to BI, the sites, investigators, or patients until the end of final database lock.



# 5.0 Analysis Populations and Stratification

#### 5.1 Analysis Populations

In this SAP, Part A refers to Week 0 to Week 16, and Part B refers to Week 16 and after.

Intent-to-Treat (ITT) Population: The ITT Population is defined as all subjects who are randomized at Week 0. ITT Population will be used for the efficacy analyses in Part A and Part B, as well as efficacy across the entire study (cross-period) for subjects who are randomized to risankizumab arms. Subjects who are randomized to placebo in Part A and do not continue into Part B will be excluded from the analysis in Part B.

ITT Population will be analyzed by treatment group as randomized.

<u>Per-Protocol (PP) Population:</u> To evaluate the impact of protocol deviations on the primary endpoint, additional efficacy analyses will be performed on a PP Population. The PP Population will include those who were most compliant with the protocol in ways that could impact the primary endpoints. Final results and the criteria for exclusion of subjects will be finalized prior to database lock.

The PP Population is defined as all subjects from the ITT Population who meet all the following criteria:

- Subjects must receive at least 75% of planned study drug injections (including dummy placebo injections) in Part A (prior to Week 16).
- Subjects must have at least one PASI assessment post-baseline.
- Inclusion Criterion 2: Subjects must have stable moderate to severe chronic plaque psoriasis at baseline:
  - Have an BSA  $\geq$  10% and
  - Have a PASI  $\geq$  12 and
  - Have an sPGA  $\geq$  3.



Final results and the criteria for exclusion of subjects will be finalized prior to the interim database lock.

PP Populations will be analyzed by treatment group as randomized.

<u>Safety Population:</u> Safety analyses will be performed on a Safety Population, comprising all randomized participants who received at least one dose of study drug in Part A. The safety analysis will be performed based on the actual treatment received at the randomization visit. Subjects who do not continue into Part B will be excluded from the Part B specific safety analysis. All safety analyses will be conducted on the Safety Population.

<u>All Risankizumab Treated (ALL RZB) Population:</u> The ALL\_RZB Population is defined as subjects who receive at least one dose of risankizumab in the study. Key safety summaries will be provided on the ALL RZB Population.

Table 1. Notation for Treatment Groups

| Population | <b>Treatment Code</b> | Definition |
|---|---|---|
| ITT/Safety | RZB_75 | Subjects who randomized to risankizumab 75 mg. |
| (Part A) | RZB_150 | Subjects who randomized to risankizumab 150 mg. |
| | PBO | Subjects who randomized to either of the two placebo arms. |
| ITT/Safety | RZB_75/RZB_75 | Subjects who randomized to risankizumab 75 mg. |
| (Part B) | RZB_150/RZB_150 | Subjects who randomized to risankizumab 150 mg. |
| | PBO/RZB_75 | Subjects who randomized to placebo and then risankizumab 75 mg entered Part B |
| | PBO/RZB_150 | Subjects who randomized to placebo and then risankizumab 150 mg entered Part B |
| ITT/Safety | RZB_75/RZB_75 | Subjects who randomized to risankizumab 75 mg. |
| (entire study) | RZB_150/RZB_150 | Subjects who randomized to risankizumab 150 mg. |
| ALL_RZB | ALL_RZB | Subjects who received at least one dose of risankizumab 75/150 mg. |



#### 5.2 Variables Used for Stratification of Randomization

Randomization will be stratified by concomitant PsA at baseline (Yes versus No) and body weight ( $\leq$  90 kg versus > 90 kg).

### 6.0 Analysis Conventions

#### **Definition of Baseline**

The last non-missing observation collected on or before the date of the first dose of study drug injection will be used as Baseline for summary of demographics and disease characteristics, safety and efficacy analyses, with the exception that:

- The last evaluation on or prior to the date of first dose of risankizumab will be used for the safety analyses in Part B among subjects randomized to placebo at Week 0, and the safety analyses in the ALL RZB Population.
- For all vital sign assessments, only assessments prior to first dose time will be considered, since vital signs are to be assessed both pre- and post-dose in some visits.

Entry of Part B is defined as the last non-missing observation collected on or before the date of the first dose of study drug in Part B for PBO/RZB\_75 and PBO/RZB\_150 arms and last non-missing observation collected on or before the date of Week 16 visit for RZB 75/RZB 75 and RZB 150/RZB 150 arms.

#### **Definition of Final Observation (Applicable to Safety Analyses)**

Final observation in Part A is defined as the last non-missing observation collected within 105 days following the last dose of study drug in Part A for those who do not enter Part B, and on or before the first dose date of study drug injection in Part B for subjects who entered Part B. For vital sign assessments, only assessments prior to the first dose of study drug injection in Part B will be included in the analysis for Part A.

Final observation for Part B is defined as the last non-missing observation collected within 105 days following the last dose in Part B.



Risankizumab M16-004 – Statistical Analysis Plan Version 1.0 – 10 Jan 2018

Final observation for the entire study analyses is defined as the last non-missing observation collected within 105 days following the last dose of study drug.

Final observation for ALL\_RZB Population is defined as the last non-missing observation collected within 105 days following the last dose of risankizumab.

# <u>Definition of Rx Days in Each Period (Days Relative to the Date of First Dose of Study Drug in Each Period)</u>

Rx Days are calculated for each time point relative to the date of first dose of study drug. They are defined as the number of days between the day of the first dose of study drug and the specific time point. Rx Days are negative values when the time point of interest is prior to the first study drug dose day. Rx Days are positive values when the time point of interest is on or after the first study drug dose day. The day of the first dose of study drug is defined as Rx Day 1, while the day prior to the first study drug dose is defined as Rx Day –1 (there is no Rx Day 0).

Rx Days for Part A and entire study will be defined relative to the date of first dose of study drug. Rx days for Part B will be defined relative to the date of the date of the first study drug injection on or after Week 16.

#### **Definition of Analysis Windows**

All time points and corresponding time windows are defined based on Rx Days. The visit schedule with accompanying details can be found in Flow Chart and Section 6.1 of the protocol.

For efficacy analyses, local tolerability, ECG, laboratory parameters, and vital sign variables, analysis windows are constructed using the following algorithm:

- Determine the nominal Rx day for each visit (e.g., Week 4 [4 weeks after Baseline visit] equals Rx Day 29).
- In order to include all post baseline data, the first post-baseline interval starts on the first day after the first dose of study drug (Rx Day 2).



- Determine the window around a specific nominal Rx day by adding or subtracting half of the interval between adjacent visits (e.g., days between Week 4 and Week 8 is 28). The threshold between adjacent visits is determined by splitting the interval evenly between the visits. If the resulting split is between Rx days, then the threshold is determined as the midpoint between the adjacent visits. If the resulting split is on an Rx day, then the threshold is determined as being between that Rx day and the Rx day prior to it (e.g., the split between Week 4 and Week 8 would be between Rx Days 43 and 44).
- If more than one assessment is included in a time window the assessment closest to the nominal day will be used. If there are two observations equidistant to the nominal day, the later one will be used in analyses. If more than one assessment is included on the same day, then the worst assessment on that day will be used in analyses, except those specified in Section 11.0.

The following analysis windows have been specified for the analysis of efficacy, laboratory parameters, and vital signs, etc. for each analysis period. In order to include all post baseline data, the first post baseline interval starts on the day after the date of first study drug injection in each period (Rx Day 2) for all efficacy variables.

For subjects who were randomized and not dosed date of randomization will be used for determining window definitions.

Table 2. Visit Windows for Analysis of PASI, Vital Signs, and Local Tolerability in Part A (ITT/PP/Safety Populations)

| Window Label | Target Day | Interval |
|--------------|------------|--------------------------|
| Baseline | 1 | ≤ 1 <sup>a</sup> |
| Week 4 | 29 | [2, 43] |
| Week 8 | 57 | [44, 71] |
| Week 12 | 85 | [72, 99] |
| Week 16 | 113 | [100, 127 <sup>b</sup> ] |

Rx Day calculated relative to first dose date of study drug. For subjects randomized but not dosed, Rx Day calculated relative to Randomization.

- a. There is no baseline for local tolerability measurements. If time is collected in vital signs, restrict to records prior to the first dose of study drug.
- b. The minimum of upper bound and the day of the first dose date in Part B (and within 105 days of last dose for safety analyses).

Table 3. Visit Windows for Analysis of Safety Laboratory Tests in Part A (Safety Population)

| Window Label | Target Day | Interval |
|--------------|------------|------------|
| Baseline | 1 | ≤ 1 |
| Week 8 | 57 | [2, 85] |
| Week 16 | 113 | [86, 141*] |

Rx Day calculated relative to first dose date of study drug.

Table 4. Visit Windows for Analysis of ECG in Part A (Safety Population)

| Window Label | Target Day | Interval |
|--------------|------------|------------|
| Baseline | 1 | ≤ 1 |
| Week 4 | 29 | [2, 71] |
| Week 16 | 113 | [72, 155*] |

Rx Day calculated relative to first dose date of study drug.

<sup>\*</sup> The minimum of upper bound, the day of the first dose date in Part B, and 105 days of last dose.

<sup>\*</sup> The minimum of upper bound, the first dose date in Part B, and the last dose + 105 days.



Table 5. Visit Windows for Analysis of sPGA, PSS, DLQI, HAQ-DI, Pain VAS, Investigator's Global Assessment VAS, Patient's Global Assessment VAS, CRP as an ACR 20 Component, SJC, and TJC in Part A (ITT Population)

| Window Label | Target Day | Interval |
|--------------|------------|-----------|
| Baseline | 1 | ≤ 1 |
| Week 16 | 113 | [2, 225*] |

Rx Day calculated relative to first dose date of study drug. For subjects randomized but not dosed, Rx Day calculated relative to Randomization.

Table 6. Visit Windows for Analysis of PASI, Vital Signs, and Local Tolerability in Part B (ITT/Safety Population)

| Window Label | Target Day | Interval |
|-----------------|------------|--------------------------|
| Entry of Part B | 1 | ≤ 1 <sup>a</sup> |
| Week 22 | 43 | [2, 64] |
| Week 28 | 85 | [65, 106] |
| Week 34 | 127 | [107, 148] |
| Week 40 | 169 | [149, 190] |
| Week 46 | 211 | [191, 232] |
| Week 52 | 253 | [233, 267] |
| Week 56 | 281 | [268, 295 <sup>b</sup> ] |

Rx Day calculated relative to the first dose date on or after Week 16 for PBO/RZB\_75 and PBO/RZB\_150 arms, and relative to the date of Week 16 visit for RZB\_75/RZB\_75 and RZB\_150/RZB\_150 arms. PASI only evaluated from Week 22 to 52. Local tolerability only evaluated from Week 22 to 40.

Subjects who enter the Open Label Extension Study 1311.31 will not have Week 56 evaluations.

<sup>\*</sup> The minimum of upper bound and the day of the first dose date in Part B.

a. If time is collected for vital sign, restrict to records prior to the first dose of study drug in Part B.

b. The minimum of upper bound and 105 days after the last dose.

Table 7. Visit Windows for Analysis of sPGA, PSS, DLQI, HAQ-DI, Pain VAS, Investigator's Global Assessment VAS, Patient's Global Assessment VAS, SJC, TJC, Laboratory Tests, and ECG in Part B (ITT/Safety Population)

| Window Label | Target Day | Interval |
|-----------------|------------|--------------------------|
| Entry of Part B | 1 | ≤ 1 |
| Week 28 | 85 | [2, 127] |
| Week 40 | 169 | [128, 211] |
| Week 52 | 253 | [212, 294 <sup>a</sup> ] |

Rx Day calculated relative to the first dose date on or after Week 16 for PBO/RZB\_75 and PBO/RZB\_150 arms, and relative to the date of Week 16 visit for RZB 75/RZB 75 and RZB 150/RZB 150 arms.

Table 8. Visit Windows for Summary of Study Drug Injections in Part A

| Window Label | Target Day | Time Window |
|--------------|------------|---------------|
| Week 0 | 1 | ≤ 1 |
| Week 4 | 29 | $[2, 57^{a}]$ |

Rx Day calculated relative to the first dose date of study drug.

Table 9. Visit Windows for Summary of Study Drug Injections in Part B

| Window Label | Target Day | Time Window |
|--------------|------------|-------------|
| Week 16 | 1 | ≤ 1 |
| Week 28 | 85 | [2, 127] |
| Week 40 | 169 | [128, 211] |

Rx Day calculated relative to the date of first dose date on or after Week 16.

#### **Definition of Missing Data Imputation**

No global imputation is taking place at the database level. Efficacy related imputations are outlined in Section 10.0. There is no imputation for missing values in the safety analyses.

a. The minimum of upper bound and 105 days after the last dose.

a. Before the first dose date on or after Week 16.



Risankizumab M16-004 – Statistical Analysis Plan Version 1.0 – 10 Jan 2018

#### **Rounding of Numeric Results**

Rounding will be performed for presentation of results. No rounding will be performed before or during analyses. The ROUND function of SAS will be used to round results.

When dichotomizing continuous variables from single observations, associated continuous variables will be rounded to 9 decimal points before applying the cutoff point to determine the response status (for example, percent change from baseline in PASI score will be rounded to 9 decimal places before comparing to 90%).

The mean and median will be rounded for presentation to 1 decimal more than the data entered into the database. The standard deviation will be rounded to 2 decimal places more than the data entered into the database. The minimum and maximum values will be presented as entered into the database.

Probabilities will be rounded to 3 decimal places before assignment of statistical significance and will be presented in rounded format. Probabilities that round to zero or are reported by SAS as zero will be presented as "< 0.001." Probabilities that round to 1 or are reported by SAS as 1 will be presented as "> 0.999."

# 7.0 Demographics, Baseline Characteristics, Medical History, and Previous/Concomitant Medications

# 7.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized for each arm and for overall of the ITT population. The number of observations, mean, standard deviation, median, minimum and maximum will be summarized for continuous variables; and treatment groups will be compared using a one-way analysis of variance (ANOVA) model with treatment as the independent factor. Categorical or discrete variables will be summarized via counts and percentages; and treatment groups will be compared using a two-sided Pearson's Chi-Square test (or an appropriate exact test if expected cell count < 5).

The following demographic and baseline parameters will be summarized.



#### **Subject Demographics**

- Sex (male, female)
- Age (years), defined as the number of years from date of birth to date of first drug
- Age (< 40 years,  $\ge 40 < 65$  years,  $\ge 65$  years)
- Body weight (kg)
- Body weight category ( $\leq$  90 kg versus > 90 kg).
- Height (cm)
- BMI  $(kg/m^2)$
- BMI (normal: < 25, over weight:  $\ge 25 < 30$ , obese:  $\ge 30$ );
- concomitant PsA at baseline

#### **General Baseline Characteristics**

- PASI (Psoriasis Area and Severity Index)
- sPGA categories
- BSA (Body Surface Area)
- PSS
- Dermatology Life Quality Index (DLQI)
- HAQ-DI (HAQ Disability Index)
- Pain VAS (Visual Analog Scale)/Patient Global Assessment (PtGA) VAS (Visual Analog Scale)
- TJC/SJC (Tender/Swollen Joints)
- Investigator's Global Assessment VAS
- Serum CRP

#### **Psoriasis and Cardiovascular History**

- Psoriatic arthritis (diagnosed, suspected, no)
- Cardiovascular Diseases (myocardial infarction, angina pectoris, transient ischemic attack, stroke, deep vein thrombosis)



Cardiovascular Risk Factors (hypertension, hyperlipidemia, diabetes mellitus, obesity)

#### **General Use**

- Smoking history (Never-smoked, Ex-smoker, Currently smokes)
- Alcohol History (Non-drinker, drinks no interference to study participation, drinks possible interference to study participation)

#### **Prior Treatment:**

- Psoriasis TNF antagonist and Other Biologic Usage History by Response to Treatment
- Psoriasis Treatment by Therapy Type (topical therapy, phototherapy, photochemotherapy, non-biologic systemic therapy, TNF antagonist, other biologic)

Physical Exam, Infection screening and Pregnancy Test will be presented in listing format.

#### 7.2 Medical History

Medical history will be summarized using body systems and condition/diagnosis as captured on the eCRF. The body systems will be presented in alphabetical order and the conditions/diagnoses will be presented in alphabetical order within each body system. The number and percentage of subjects with a particular condition/diagnosis will be summarized for each treatment arm. Subjects reporting more than one condition/diagnosis within a body system will be counted only once for that body system.

#### 7.3 Previous Treatment and Concomitant Medications

Prior and concomitant medications will be summarized by generic name. A prior medication is defined as any medication taken at the time of entry into the study and prior



to the first dose of study drug. A concomitant medication is defined as any medication that started prior to the first dose of study drug and continued to be taken after the first dose of study drug or any medication that started after the first dose of study drug, but not after the last dose of study drug plus 21 days. The number and percentage of subjects who had taken medications will be summarized by generic drug name assigned by the World Health Organization (WHO) for both prior and concomitant medications.

#### 7.4 Protocol Deviations

Number and percentage of subjects who reported at least one of the following protocol deviation categories will be provided.

- Subject entered into the study even though she/he did not satisfy entry criteria
- Subject who developed withdrawal criteria during the study and was not withdrawn
- Subject who received wrong treatment or incorrect dose
- Subject who received excluded or prohibited concomitant treatment

# 8.0 Patient Disposition

The number of subjects for each of the following categories will be summarized, for overall and for each treatment group in the ITT population:

- Number of subjects randomized
- Number of subjects treated
- Number of subjects who completed the study
- Number of subjects who discontinued the study drug
- Number of subjects who prematurely discontinued study

In addition, the reasons for premature discontinuation will be summarized with frequencies and percentages.



In addition to patient disposition, number of screening failures and reasons for screening failure will also be summarized among all screened subjects in a subject screening status table.

The summaries will be provided for Part A and Part B.

# 9.0 Study Drug Exposure and Compliance

Summary of study drug treatment duration and compliance will be provided for each treatment arm in each treatment period under the ITT Population.

Study drug treatment duration (days) will be summarized using the sample size, mean, standard deviation, minimum, median and maximum. In addition cumulative exposure of RZB (including total patient years) will also be summarized in the ALL\_RZB Population. Study drug treatment duration will be summarized as follows:

#### **Study Drug Exposure (in Days) in Each Period:**

#### Part A:

- For subjects who did not continue into Part B:
  - Date of last injection in Part A Date of first injection in Part A + 84 days.
- For subjects who continued into Part B:

Minimum of

- Date of first injection in Part B Date of first injection in Part A
- Date of last injection in Part A Date of first injection in Part A + 84 days.

#### Part B:

Date of last injection in Part B – Date of first injection in Part B + 84 days.

#### **ALL RZB:**

For study drug exposure during the administration of risankizumab in the ALL\_RZB Population:



Date of last injection of risankizumab – Date of first injection of risankizumab + 84 days.

A data cutoff date (December 15, 2017) will be applied during the interim analysis, and the duration of study drug exposure will be defined up to this cutoff date.

#### **Compliance**

There will be a summary of the number of subjects receiving study drug and dose at each study drug administration visit. This will be repeated on the cumulative number of doses.

When computing compliance at each study drug administration visit, the denominator will include all subjects in each analysis population who have not prematurely discontinued the study drug prior to the scheduled study drug injection. Subjects who have prematurely discontinued the study drug but have not prematurely discontinued the study are not used in the denominator.

# 10.0 Efficacy Analysis

#### 10.1 General Considerations

When the last patient completes the Week 28 visit, the Primary Analysis will be performed including all efficacy endpoints pertaining to Part A. This is the only and final analysis for these endpoints, hence no alpha adjustment is required. For this primary analysis, all endpoints will be analysed up to Week 28, with the following exception:

 Categorical endpoints related to PASI and sPGA, using the LOCF method, will be analysed up to the last visit that at least one subject has observed PASI and sPGA measurements, respectively.

The treatment effect will be evaluated based on a two-sided significance level of 0.05 (when rounded to three decimal places).

The ITT population will be used for the analyses of efficacy endpoints. The following treatment periods will be analyzed:

- Part A (up to Week 16)
- Part B (Week 16 and after)

Time-to-event analysis will be performed across the entire study for subjects who are randomized to risankizumab or placebo arms in addition to the analyses in Part A.

Primary variable will also be analyzed for the per-protocol populations using primary approach to handle missing data as described in Section 10.1.4.

Subjects' actual Concomitant PsA at baseline (Yes: Diagnosed or Suspected; versus: No) and body weight ( $\leq 90 \text{ kg versus} > 90 \text{ kg}$ ) will be used as the strata in the stratified analyses.

# 10.1.1 Analyses of Categorical Variables

For categorical variables, frequencies and percentages will be summarized. Treatment comparison will be conducted using a Cochran-Mantel-Haenszel (CMH) test with stratification factors as strata for the analysis. The CMH test will use weights proposed by Greenland & Robins, which is calculated as follows:

$$\hat{\delta}_{MH} = rac{\sum_{i=1}^{u} w_i \cdot \hat{\delta}_i}{\sum_{i=1}^{u} w_i}$$
 , where

$$\hat{\delta}_i = \frac{x_i}{n_i} - \frac{y_i}{m_i}$$
 denotes the risk difference in stratum  $i, i = 1, \cdots, u$ 

$$w_i = \frac{n_i \cdot m_i}{n_i + m_i}$$
 denotes the weight of stratum  $i, i = 1, \dots, u$ 

 $x_i$  denotes the number of subjects with event in treatment<sub>1</sub> in stratum i,  $i=1,\cdots,u$   $y_i$  denotes the number of subjects with event in treatment<sub>2</sub> in stratum i,  $i=1,\cdots,u$ 

 $n_i$  denotes the number of subjects on treatment<sub>1</sub>in stratum i,  $i=1,\cdots,u$   $m_i$  denotes the number of subjects on treatment<sub>2</sub>in stratum i,  $i=1,\cdots,u$ 

The estimated variance of  $\hat{\delta}_{MH}$  is calculated as:

$$\widehat{var}(\hat{\delta}_{MH}) = \frac{\sum_{i=1}^{u} L_i}{(\sum_{i=1}^{u} w_i)^2}$$

where 
$$L_i = \frac{x_i(n_i - x_i) m_i^3 + y_i(m_i - y_i) n_i^3}{n_i \cdot m_i \cdot (n_i + m_i)^2}$$
,  $i = 1, \dots, u$ 

Assuming a normal distribution of  $\hat{\delta}_{MH}$ , an approximate 95% CI is given as follows, where  $z_{0.975}$  is the 97.5% quantile of the standard normal distribution:

$$CI = \left[ \hat{\delta}_{MH} \pm z_{0.975} \cdot \sqrt{\widehat{var}(\hat{\delta}_{MH})} \right]$$

Also, the approximate p-value can be calculated using the following:

pvalue = 
$$2 \cdot \Pr \left[ Z > \left| \frac{\hat{\delta}_{MH}}{\sqrt{\widehat{var}(\hat{\delta}_{MH})}} \right| \right]$$
, where  $Z \sim N(0, 1)$ 

If there is a stratum for a treatment group that has 0 subjects in any cell in the contingency table, all cells from the stratum will be added by 0.1 in order to prevent dividing by 0 in the above equations, as suggested in Greenland & Robins.

# 10.1.2 Analyses of Continuous Variables

Change from baseline in PSS will be analyzed by stratified van Elteren test. For other continuous variables, the model based mean and standard error will be presented. The Baseline and visit means will also be presented for each treatment group for subjects who



have both Baseline and post Baseline visit values. The treatment groups will be compared using ANCOVA with treatment group, Baseline value, and stratification factors in the model.

### 10.1.3 Analyses of Time-to-Event Variables

Time-to-event analysis will be done for RZB\_75, RZB\_150, PBO treatment arms for Part A, and all RZB\_75/ RZB\_75, RZB\_150/ RZB\_150 treatment arms for the entire study.

For the time to first achievement of Endpoint, the time to event will be calculated as:

- Time to first achievement (with observed event) = [date of first achievement] [date of first study drug] + 1
- If a subject never attains an endpoint, then that subject's time to first achievement will be censored at the last visit where variable was measured. Censoring will be done within Part A for the analyses in Part A, and over the entire study for cross-period analyses. For example, if the first time a PASI 90 response is achieved in Part B, then PASI 90 will be censored for Part A analysis only.

Time to loss of response will be evaluated from the time of achievement of the same endpoint, and defined using the following algorithm:

- Never attains Endpoint (Failure at time 0)
- After achieving Endpoint, subjects will be a considered loss of response if they subsequently lost the response or discontinue from the study due to AE of "Worsening of disease under study."
- Subjects will be censored at their last assessment if they do not lose the
  endpoint or discontinue from the study due to reasons other than AE of
  "Worsening of disease under study." Time to failure will be calculated starting
  from date of first achievement of the endpoint.



Time to event will be analyzed using Kaplan-Meier estimates for each treatment group. Treatments comparisons will be performed using stratified Log-rank test.

# 10.1.4 Missing Data Imputations

Missing data will be imputed using the following methods for the efficacy analyses:

- Non-Responder Imputation (NRI): The NRI analysis will categorize any subject who has missing value at a specific visit as non-responder for that visit. The only exception is when if the subject is a responder both before and after this specific visit window, then the subject will be categorized as a responder for the visit. The NRI will be the primary approach in the analysis of categorical variables. Of note, this before- and after-window imputation will utilize visits across Part A and B for the risankizumab arms.
- Last Observation Carried Forward (LOCF): The LOCF analyses will use the completed evaluation from the previous visit for efficacy measures assessed to impute missing data at later visits. For observations in RZB\_75/RZB\_75, and RZB\_150/RZB\_150 arms in Part B, LOCF is continued across Part A and Part B. LOCF will be applied to the observations in PBO/RZB\_75, and PBO/RZB\_150 arms within the analysis period. Baseline values will not be carried forward. LOCF will be the primary approach in the analyses of continuous variables, and the secondary approach in the analyses of categorical variables.
- As-observed: The as-observed analysis will not impute values for missing evaluations, and thus a subject who does not have an evaluation on a scheduled visit will be excluded from the as observed analysis for that visit. As-observed analysis will be the secondary approach in the analysis of continuous variables.
- Multiple Imputation (MI): The MI will be used as sensitivity approach to impute missing data in primary endpoints. The variables to be included in the imputation model are listed below. If MI is not applicable due to the nature of our data (e.g., MCMC algorithm does not converge), logistic regression or mixed effect model repeat measurement (MMRM) methods will be applied as sensitivity approach, whichever applicable.



The Multiple Imputation analysis will be carried out in three steps.

- Imputation of missing data. The imputation will be generated for each efficacy endpoint measurement. The variables to be included in the imputation model are: concomitant disease of Baseline disease severity (PASI and sPGA), Baseline weight, treatment group, Concomitant PsA at baseline (Yes: Diagnosed or Suspected; versus: No), and measurements at each visit from randomization up to the end of the analysis period. For each endpoint, 20 'complete' datasets will be generated using SAS PROC MI. The imputed post-baseline measurements will be rounded to the same precision as the observed data before the determination of responder status (e.g., PASI90).
- Analysis of imputed data sets. A CMH test, stratified by stratification factors, will be used to analyze categorical endpoints in each imputed dataset.
- Synthesis of imputation and analysis results. SAS PROC MIANALYZE will be used to generate the final inferences of the risk difference between treatment groups.

Of note, subjects who discontinued due to AE of "worsening of disease under study" will be counted as non-responders in all subsequent visits in the NRI and MI analyses, and will have their last observation prior to discontinuation carried forward in the LOCF analyses. For Observations in RZB\_75/RZB\_75, and RZB\_150/RZB\_150 arms in Part B, LOCF is continued across Part A and Part B. LOCF will not carry forward from Period A to Period B for PBO/RZB 75, and PBO/RZB 150 arms.

#### 10.1.5 Analysis of Psoriasis Symptoms Scale (PSS)

The 4-item PSS was designed to measure patient-reported psoriasis symptoms. Subjects are requested to rate the severity of each of their symptoms related to pain, redness, itching, and burning, in the last 24 hours from "0 = none" to "4 = very severe," with total scores, which is the sum of the four item responses, ranging from 0 to 16 with higher scores indicating worse symptoms. If one or more of the four items are missing then the total score for that day will be set to missing.



proc freq data = indata;

PSS will be completed on Day 1 and the Week 16 visit in Part A. Total Score from Day 1 will be used as the baseline value. Change from baseline in PSS will be analyzed by the van Elteren test between the risankizumab arms and placebo arm using the stratification factors of Concomitant PsA at baseline (Yes: Diagnosed or Suspected; versus: No) and body weight ( $\leq$  90 kg versus > 90 kg). An example of the SAS code for this is as follows:

```
tables strata * treatmnt * aval1 / cmh2 scores=modridit noprint;
```

where "strata" is numbered 1-4 based on the row order, "treatment" is dichotomous (Arm A or Arm B), and "aval1" is the PSS change from baseline at Week 16. In the output from this code, the p-value is the "Prob" for statistic 2- "Row Mean Scores Differ"

PSS will be completed by the subject during clinic visits at Week 28, Week 40 and Week 52 in Part B. The PSS change from baseline will be summarized for these visits for each treatment arm

In addition to the PSS total score, the four individual components, pain, redness, itching, and burning, will be analyzed using the same methodology.

# 10.2 Primary Efficacy Analysis

The primary hypotheses is that either risankizumab 150 mg or risankizumab 75 mg is superior to placebo in achieving  $\geq 90\%$  reduction from baseline in the PASI score (PASI 90) at Week 16 in participants with moderate to severe chronic plaque psoriasis.

In order to maintain the full significant level of 5%, the following null hypotheses will be tested in rank order, with two-sided alpha level 0.05.

1. Risankizumab 150 mg is not different from placebo with respect to PASI 90 response at Week 16



2. Risankizumab 75 mg is not different from placebo with respect to PASI 90 response at Week 16

The difference in proportion of subjects achieving PASI 90 between treatment arms will be estimated and tested using the Cochran-Mantel-Haenszel risk difference estimate stratified by the stratification factors of Concomitant PsA at baseline (Yes: Diagnosed or Suspected; versus: No) and body weight (≤ 90 kg versus > 90 kg).

The primary analysis will be carried out in the ITT Population and the PP Population. Non-responder imputation will be used as the primary approach for missing values. LOCF and MI will be performed as sensitivity analyses.

# 10.3 Secondary Efficacy Analyses

Secondary endpoints will be analysed in the ITT Population. The same methods as discussed for the primary analyses will be used to analyze all binary secondary endpoint at Week 16.

Secondary endpoints for Week 52 will be summarized descriptively.

Secondary Efficacy Endpoints are:

- Achievement of PASI 90 at Week 52
- Achievement of an sPGA score of clear or almost clear at Week 16
- Achievement of an sPGA score of clear or almost clear at Week 52
- Achievement of ≥ 75% reduction from baseline PASI score (PASI 75) at Week 16
- Achievement of PASI 75 at Week 52
- Achievement of 100% reduction from baseline PASI score (PASI 100) at Week 16
- Achievement of PASI 100 at Week 52



- Achievement of an American College of Rheumatology (ACR) 20 response at Week 16, among subjects with confirmed diagnosis of PsA using CASPAR criteria and with baseline total TJC and SJC counts ≥ 3 at selected study sites
- Achievement of an ACR 20 at Week 52, among subjects with confirmed diagnosis of PsA using CASPAR criteria and with baseline total TJC and SJC counts ≥ 3 at selected study sites

#### 10.3.1 Further Efficacy Analysis

Further exploratory endpoints below will be analyzed among the ITT Population at all visits collected:

- Achievement of PASI 50/75/90/100
- Achievement of sPGA of clear and sPGA of clear or almost clear
- Time until the first achievement of PASI 50, PASI 75, PASI 90, PASI 100, sPGA of clear and sPGA of clear or almost clear
- Time until loss of PASI 75, PASI 90, PASI 100, sPGA of clear and sPGA of clear or almost clear response
- Change from baseline in PASI score
- Percent change from baseline in PASI
- Achievement of absolute PASI of < 3
- Change from baseline in psoriasis symptoms evaluated using the total score on the Psoriasis Symptoms Scale (PSS)
- Achievement of a Dermatology Life Quality Index (DLQI) score of 0 or 1
- Achievement of total score on the PSS of 0
- Change from baseline in DLQI
- Change from baseline in HAQ-DI, among subjects with confirmed diagnosis of PsA using CASPAR criteria and with baseline total TJC and SJC counts ≥ 3 at selected study sites
- Change from baseline in Pain VAS, among subjects with confirmed diagnosis of PsA using CASPAR criteria and with baseline total TJC and SJC counts ≥ 3 at selected study sites



- Change from baseline in Patient's Global Assessment VAS, among subjects with confirmed diagnosis of PsA using CASPAR criteria and with baseline total TJC and SJC counts ≥ 3 at selected study sites
- Change from baseline in Investigator's Global Assessment VAS, among subjects with confirmed diagnosis of PsA using CASPAR criteria and with baseline total TJC and SJC counts ≥ 3 at selected study sites
- Achievement of an ACR 20, among subjects with confirmed diagnosis of PsA using CASPAR criteria and with baseline total TJC and SJC counts ≥ 3 at selected study sites
- Investigator's global assessment among subjects with confirmed diagnosis of PsA using CASPAR criteria and with baseline total TJC and SJC counts ≥ 3 at selected study sites
- Change from baseline in CRP, among subjects with confirmed diagnosis of PsA using CASPAR criteria and with baseline total TJC and SJC counts ≥ 3 at selected study sites
- Change from baseline in TJC and SJC, among subjects with confirmed diagnosis of PsA using CASPAR criteria and with baseline total TJC and SJC counts ≥ 3 at selected study sites

In addition, the proportion of subjects achieving PASI 90, PASI 100, sPGA of clear, and sPGA of clear or almost clear at each visit in Part B will be summarized among those who had PASI 90, PASI 100, sPGA of clear, and sPGA of clear or almost clear, respectively, at the entry of Part B.

#### 10.4 Handling of Multiplicity

The statistical comparisons for the primary efficacy will be carried out in the hierarchical order:

- 1. The risankizumab 150 mg groups vs the placebo group.
- 2. The risankizumab 75 mg groups vs the placebo group.



The statistically significant results (p-value  $\leq 0.05$ ) for the comparison in the higher rank are necessary to initiate the testing of the next comparison in the lower rank. Since a step-down procedure is used, each comparison will be tested at a significance level of 0.05 and overall alpha level of 0.05 will be preserved.

# 10.5 Efficacy Subgroup Analysis

To evaluate the consistency of the efficacy on the primary endpoint of PASI 90 at Week 16 over demographic and other baseline characteristics, summaries and analyses will be performed for the following subgroups.

- Age ( $< 40 \text{ years}, \ge 40 < 65 \text{ years}, \ge 65 \text{ years}$ )
- Sex (male, female)
- Smoking (current, ex or never)
- BMI (normal: < 25, over weight:  $\ge 25 < 30$ , obese:  $\ge 30$ );
- Body weight ( $\leq 90 \text{ kg versus} > 90 \text{ kg}$ )
- Body weight (≤ median versus > median)
- Baseline PASI score (by median);
- Baseline sPGA (3, 4)
- concomitant PsA at baseline (Yes: baseline total TJC and SJC counts  $\geq 3$  versus No: otherwise) among the subjects at the selected sites
- Psoriasis Therapy History (Phototherapy or Photochemotherapy, TNF Antagonist, Other biologics, Non-biologic systemic therapy, All biologics, Naïve to all)

# 11.0 Safety Analysis

#### 11.1 General Considerations

Safety analyses will include adverse events, laboratory, local tolerability, ECG, and vital sign measurements. Safety summaries will be provided using the safety population as defined in Section 5.1. Pairwise comparisons of risankizumab vs placebo will be



performed in the Safety Population. Continuous variables will be analyzed using one-way ANOVA and categorical variables will be analyzed using Fisher's exact test. For analyses of AEs, only P values  $\leq 0.100$ , when rounded to three digits, will be presented.

Missing safety evaluations will not be imputed.

#### 11.2 Analysis of Adverse Events

#### 11.2.1 Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as any event with an onset that is after the first dose of study drug and with an onset date within 105 days after the last dose of study drug in the analysis period, or prior to the first dose in the subsequent period for subjects who entered in to the subsequent period. Events where the onset date is the same as the study drug start date are assumed to be treatment-emergent, unless the adverse event start time is prior to the study drug start time. If an incomplete onset date is collected for an adverse event, the event will be assumed to be treatment-emergent unless there is other evidence that confirms that the event is not treatment-emergent (e.g., the event end date is prior to the study drug start date).

The data cutoff date (December 15, 2017) will be applied to TEAEs during the interim analysis, in accordance to the duration of study drug exposure defined up to this cutoff date.

#### Summary tables will be presented as follows:

#### 1. Adverse Event Overview

The number and percentage of subjects experiencing treatment-emergent adverse events will be summarized for the following adverse event categories.

- Any AE
- Any AE that was assessed as related to study drug by the investigator
- Any severe AE
- Any serious AE (SAE)



- Any SAE that was assessed as related to study drug by the investigator
- Any AE leading to discontinuation of study drug.
- Any AE leading to death.
- Any deaths
- Areas of Safety Interest

#### 2. Adverse Events by System Organ Class and Preferred Term

TEAEs will be summarized and presented using primary Medical Dictionary for Regulatory Activities (MedDRA) system organ classes (SOCs) and preferred terms (PTs). The SOCs will be presented in alphabetical order, and the PTs will be presented in alphabetical order within each SOC.

Subjects reporting more than one adverse event for a given MedDRA preferred term will be counted only once for that term (most severe incident for the severity tables and most related incident for the relationship tables). Subjects reporting more than one type of adverse event within a SOC will be counted only once for that SOC. Subjects reporting more than one type of adverse event will be counted only once in the overall total.

In addition, the number and percentage of adverse events with causal relationship between the events and the study drug will be summarized using the same conventions described above.

#### 3. Adverse Events by Maximum Severity

The severity grading of AEs follows Rheumatology Common Toxicity Criteria (RCTC).

- Grade 1 mild
- Grade 2 moderate
- Grade 3 severe
- Grade 4 life threatening

Adverse events will be summarized by maximum severity. If a subject has an adverse event with unknown severity, then the subject will be counted in the



severity category of "unknown," even if the subject has another occurrence of the same event with a severity present. The only exception is if the subject has another occurrence of the same adverse event with the most extreme severity (life threatening). In this case, the subject will be counted under the "life threatening" category.

#### 4. Adverse Events by Maximum Relationship

Adverse events will be summarized by maximum relationship to study drug, as assessed by the investigator. Relationship of an AE to study drug is assessed by the investigator and collected in the CRF as 'Yes' or 'No.' If a subject has an adverse event with unknown relationship, the subject will be counted in the relationship category of "unknown," even if the subject has another occurrence of the same event with a relationship of "No." If the subject has another occurrence of the same adverse event with a relationship assessment of "Yes," the subject will be counted under the "yes" category.

A listing of all pretreatment (i.e., events start prior to the first study drug injection) serious adverse events will be provided.

The following tables are planned.

#### Treatment-emergent adverse events will be summarized as follows:

- Grouped by SOC and PT
- Grouped by SOC, PT and maximum relationship to study drug
- Grouped by SOC, PT and maximum severity

#### **Treatment-emergent SAEs will be summarized as follows:**

- Grouped by SOC and PT
- A by-subject listing will be provided



#### Pre-treatment SAEs will be summarized as follows:

• A by-subject listing will be provided

# Treatment-emergent adverse events leading to death or premature discontinuation of study drug will be summarized as follows:

- Grouped by SOC and PT
- Separate listings by subject for deaths and premature terminations of study drug due to adverse events will be provided.

#### Treatment-emergent areas of safety interest will be summarized as follows:

- Grouped by SOC and PT
- A listing by subject will be provided.

#### **Areas of Safety Interest**

Areas of Safety Interest groupings are listed in Table 10. These events are of interest due to a higher rate in the moderate to severe psoriasis population, or of interest for all immunoglobulin products or products in general.

The final list will be based on the most updated final version of risankizumab Product Safety Statistical Analysis Plan, which is consistent to the most updated risankizumab Risk Management Plan.



# Table 10. Areas of Safety Interest

| ASI Grouping | Categories<br>(ASI) | Search Criteria | Terms to Display | Include<br>in AE<br>Overview<br>(Y/N) |
|---|---|---|---|---|
| Adjudicated CV<br>Events | MACE | Adjudicated events | Display underlined terms defined by the following adjudicated terms: • CV Death which includes CETERM values: Fatal CV, Fatal PE, Fatal Non- Cardiac/Non-Neuro Arterial Thrombosis/Thromboembol ism, Undetermined Death, Not assessable death (cardiac/neuro/thrombotic), Fatal Stroke • Myocardial infarction • Stroke | Y |
| | Extended<br>MACE | Adjudicated events | Display underlined terms from MACE and underlined terms below: • Hospitalization for Unstable Angina • Coronary Revascularization Procedures | N |


Table 10. Areas of Safety Interest (Continued)

| ASI Grouping | Categories<br>(ASI) | Search Criteria | Terms to Display | Include<br>in AE<br>Overview<br>(Y/N) |
|---|---|---|---|---|
| Adjudicated CV<br>Events<br>(continued) | Other CV events | Adjudicated events | Display underlined terms defined by the following adjudicated terms: • Thrombotic events which includes CETERM values: Deep Vein Thrombosis, TIA, Pulmonary Embolism, Non-fatal Non- Cardiac/Non-Neurological Arterial Thrombosis/ Thromboembolism, Other Venous Thrombosis, specified (non-fatal) • Cardiac arrhythmia which includes CETERM of: Clinically Significant Arrhythmia • Congestive heart failure which includes CETERM of Heart Failure • Hypertensive emergency | N |
| Serious<br>infections, TB,<br>fungal and<br>opportunistic<br>infections<br>(including<br>herpes zoster) | Serious<br>infections | Serious PTs of<br>the CMQ<br>(company<br>MedDRA query)<br>Infections<br>(CMQ 80000018) | PTs | Y |
| | ТВ | Tuberculosis (including Investigations) CMQ (code 80000033) | PTs | Y |
| | Opportunistic infections | Opportunistic infections CMQ (code 80000073) | PTs | N |



Table 10. Areas of Safety Interest (Continued)

| ASI Grouping | Categories<br>(ASI) | Search Criteria | Terms to Display | Include<br>in AE<br>Overview<br>(Y/N) |
|---|---|---|---|---|
| Serious infections, TB, fungal and | Fungal infections | Fungal infections<br>CMQ<br>(code 80000063) | PTs | N |
| opportunistic<br>infections<br>(including<br>herpes zoster)<br>(continued) | Herpes Zoster | Herpes zoster<br>CMQ<br>(code 80000175) | PTs | N |
| Malignancies | All possible malignancies | Narrow –<br>Malignancies<br>(SMQ 20000090) | PTs | N |
| | Malignant<br>Tumours | Narrow –<br>Malignant<br>tumours<br>(SMQ 20000194) | PTs | Y |
| | Non-melanoma<br>skin cancer<br>(NMSC) | Broad – Skin<br>malignant<br>tumours<br>(SMQ 20000204)<br>excluding terms<br>identified by the<br>Melanoma CMQ<br>(code 80000119) | PTs | N |
| | Malignant<br>Tumours<br>excluding<br>NMSC | 'Malignant Tumours excluding NMSC' is identified by the 'Malignant Tumours' search excluding terms identified by the 'Non-melanoma skin cancer (NMSC) search. | PTs | Y |



Table 10. Areas of Safety Interest (Continued)

| ASI Grouping | Categories<br>(ASI) | Search Criteria | Terms to Display | Include<br>in AE<br>Overview<br>(Y/N) |
|---|---|---|---|---|
| Hypersensitivity<br>Reaction | Hypersensitivity | Narrow –<br>Hypersensitivity<br>(SMQ 20000214) | PTs | Y –<br>serious<br>events<br>only |
| | Anaphylactic<br>Reaction | Narrow –<br>Anaphylactic<br>reaction<br>(SMQ 20000021) | PTs | N |
| Hepatic Events | Hepatic Events | Broad – Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions (SMQ 20000013) Broad – Hepatitis, non-infectious (SMQ 20000010) Broad – Cholestasis and jaundice of hepatic origin (SMQ 20000009) Broad – Liver related investigations, signs and symptoms (SMQ 20000008) Narrow – Liver-related coagulation and bleeding disturbances (SMQ 20000015) | PTs | N |



#### Adverse Event per 100 Patient-Years of Exposure

AEs occurring during the entire study will be presented by event rate per 100 patient years. These will be presented for any TEAEs, serious adverse events, Areas of Safety Interest.

AEs per 100 patient-years of exposure is defined as the number of AEs divided by the total exposure in 100 patient-years. Note that one event per preferred term per day per subject will be counted in the calculation of the number of AEs (i.e., a preferred term will not be counted twice on the same day for the same subject). See the calculation method below.

$$100 \times \frac{\text{Number of TEAEs}}{\text{Total Patient Years}}$$

where total patient years is defined as the sum of the study drug exposure (defined as date of last dose – date of first dose + 105 days (5 half-lives)) of all subjects normalized by 365.25, and rounded to one decimal place.

# 11.2.2 SAEs (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation

Deaths and all SAEs will be presented in listing format. In addition, SAEs will be summarized by System Organ Class and MedDRA Preferred Term.

#### 11.2.3 Safety Subgroup Analysis

The AE overview and AE by SOC and preferred term in each period will also be analyzed with respect to the actual values of:

- concomitant PsA at baseline (Yes: baseline total TJC and SJC counts  $\geq 3$  versus No: otherwise) among the subjects at the selected sites
- Dichotomous body weight ( $\leq 90 \text{ kg versus} > 90 \text{ kg}$ )
- Dichotomous body weight (≤ median versus > median)



## 11.3 Analysis of Laboratory Data

For the assessments of laboratory data, values observed more than 105 days after the last dose of study drug will be excluded.

Listing and descriptive statistics of laboratory values over time, change from baseline, and extreme abnormal value on treatment will be provided. Extreme abnormal value is the value which is most significantly away from the reference range. Frequency of subjects with transitions relative to reference range and listing of subjects with significant abnormal laboratory values will be presented as well.

## 11.3.1 Variables and Criteria Defining Abnormality

Clinical laboratory tests performed by central laboratory service provider are listed below.



Table 11. Clinical Laboratory Tests

| Category | Test Name | |
|-----------------------|---------------------------------------------|---|
| Haematology | Hematocrit (Hct) | |
| | Hemoglobin (Hb) | |
| | Glycosylated Hbc (HbA1c) | |
| | White Blood Cells/Leukocytes | |
| | Platelet Count/Thrombocytes | |
| Diff. Automatic | Neutrophils (relative and absolute count) | |
| | Eosinophils (relative and absolute count) | |
| | Lymphocytes (relative and absolute count) | |
| Enzymes | AST (GOT) | |
| | ALT (GPT) | |
| | Alkaline Phosphatase (AP) | |
| | Creatine Kinase (CPK) | |
| | Gamma-Glutamyl Transferase (GGT/γ-GT) | |
| | Lactic Dehydrogenase (LDH) | |
| | Amylase | |
| | Lipase | |
| Electrolytes | Calcium | |
| | Sodium | |
| | Potassium | |
| Substrates | Glucose | |
| | BUN | |
| | Uric acid | |
| | Creatinine | |
| | eGFR (estimated by CKD-EPI formula) | |
| | Bilirubin Total | |
| | Albumin | |
| | C-Reactive Protein (CRP) (high sensitivity) | |
| | Cholesterol, total | |
| | Triglycerides | ļ |
| | LDL-Cholesterol | ļ |
| | HDL-Cholesterol | |
| Urinalysis (dipstick) | Urine Glucose | |



#### 11.3.2 Statistical Methods

All analyses will be conducted in the Safety Population. Table for potentially clinically important lab values will also be summarized in the ALL\_RZB Population.

#### **Analysis of Continuous Laboratory Parameters**

Though the protocol indicates utilizing the Rheumatology Common Toxicity Criteria (RCTC) scale for grading laboratory values, given that the NCI National Cancer Institute Common Toxicity Criteria for Adverse Event (CTCAE) scale includes a more comprehensive list of laboratory values; therefore, the lab analyses based on the NCI CTCAE scale will be presented. Change from Baseline to each scheduled visit and to the final value in continuous laboratory parameters will be summarized with the mean, standard deviation and median. The Baseline and visit/final value means will also be presented for subjects who have both the Baseline and visit/final values (see Section 6.0 for the definition of Baseline and final values). If there are multiple post-baseline measurements on the same day, the average value will be used.

#### **Shift Tables**

Shift tables for changes from Baseline according to the normal range will be provided for each hematology and clinical chemistry parameter. Shifts from Baseline to the following endpoints will be considered: minimum value, maximum value and final value. Categories of "low or normal" and "high or normal" will be included at Baseline in addition to the categories of "low," "normal," "high" and "missing." If there are multiple measurements on the same day, the last value will be used.

#### **Potentially Clinically Important Laboratory Values**

Frequencies and percentages of subjects with post Baseline lab values meeting the following criteria will be summarized. Of note, a post baseline value must be more extreme than the baseline value to be considered a potentially clinically important finding.



Table 12. Criteria for Potentially Clinically Important Chemistry Values

| | | Definition of Potentially Clinically Important Curren<br>(Version 4) NCI CTCAE Grade 3 or Greater | |
|---|---|---|---|
| <b>Chemistry Variables</b> | Units | Very Low | Very High |
| TBL | mcmol/L | | > 3.0 × ULN |
| SGOT/AST | U/L | | $> 5.0 \times ULN$ |
| SGPT/ALT | U/L | | $> 5.0 \times ULN$ |
| Albumin | g/L | < 20 | |
| Glucose | mmol/L | < 2.2 | > 13.9 |
| Triglycerides | mmol/L | | > 5.7 |
| Creatinine | mcmol/L | | $> 3.0 \times ULN$ |
| Sodium | mmol/L | < 130 | > 155 |
| Potassium | mmol/L | < 3.0 | > 6.0 |
| Calcium | mmol/L | < 1.75 | > 3.1 |
| CPK | U/L | | $> 5.0 \times ULN$ |
| Total Cholesterol | mmol/L | | > 10.34 |
| GGT | | | $> 5.0 \times ULN$ |
| ALP | | | $> 5.0 \times ULN$ |
| Lipase | | | $> 5.0 \times ULN$ |
| Amylase | | | $> 5.0 \times ULN$ |

Table 13. Criteria for Potentially Clinically Important Hematology Values

| | | Definition of Potentially Clinically Important Current<br>(Version 4) Grade 3 or Greater |
|---|---|---|
| Hematology Variables | Units | Very Low |
| Hemoglobin | g/dL | < 8.0 |
| Platelets count | $10^{9}/L$ | < 50.0 |
| WBC count | $10^{9}/L$ | < 2.0 |
| Neutrophils | $10^{9}/L$ | < 1.0 |
| Lymphocytes | $10^{9}/L$ | < 0.5 |

A separate listing will be provided that presents all of the subjects and values that are NCI CTCAE toxicity grade 3 or above. For each of these subjects, the whole course of the

respective parameter will be listed. The NCI CTCAE grading is shown in Table 14 below:

Table 14. NCI CTCAE Grading

| Test | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| SGPT/ALT increased | $>$ ULN $-3.0 \times$ ULN | $> 3.0 - 5.0 \times ULN$ | $> 5.0 - 20.0 \times ULN$ | > 20.0 × ULN |
| SGOT/AST increased | $>$ ULN $-3.0 \times$ ULN | $> 3.0 - 5.0 \times ULN$ | $> 5.0 - 20.0 \times ULN$ | > 20.0 × ULN |
| GGT increased | $>$ ULN $-2.5 \times$ ULN | $> 2.5 - 5.0 \times ULN$ | $> 5.0 - 20.0 \times ULN$ | $> 20.0 \times ULN$ |
| ALP increased | $>$ ULN $-3.0 \times$ ULN | $> 3.0 - 5.0 \times ULN$ | $> 5.0 - 20.0 \times ULN$ | $>20.0\times ULN$ |
| TBL increased | $>$ ULN $-1.5 \times$ ULN | $> 1.5 - 3.0 \times ULN$ | $> 3.0 - 10.0 \times ULN$ | $> 10.0 \times ULN$ |
| Creatinine increased | $>$ ULN $-1.5 \times$ ULN | $> 1.5 - 3.0 \times ULN$ | $> 3.0 - 6.0 \times ULN$ | > 6.0 × ULN |
| CPK increased | $>$ ULN $-2.5 \times$ ULN | $> 2.5 - 5.0 \times ULN$ | $> 5.0 - 10.0 \times ULN$ | $> 10.0 \times ULN$ |
| Hemoglobin decreased | < LLN – 100.0 g/L | < 100.0 – 80.0 g/L | < 80.0 | |
| Neutrophil count decreased | $< LLN - 1.5 \times 10^9 / L$ | $< 1.5 - 1.0 \times 10^9 / L$ | $< 1.0 - 0.5 \times 10^9 / L$ | $<0.5\times10^9/L$ |
| WBC decreased | $< LLN - 3.0 \times 10^9/L$ | $< 3.0 - 2.0 \times 10^9 / L$ | $< 2.0 - 1.0 \times 10^9 / L$ | $< 1.0 \times 10^{9}/L$ |
| Lymphocyte count decreased | $< LLN - 0.8 \times 10^9/L$ | $< 0.8 - 0.5 \times 10^9 / L$ | $< 0.5 - 0.2 \times 10^9 / L$ | $<0.2\times10^9/L$ |

If there are multiple post-baseline measurements on the same day, the worst value will be used.

#### **Liver Function Tests**

Additional summaries will be presented for liver function tests including ALT or serum glutamic-pyruvic transaminase (SGPT), AST or serum glutamic-oxaloacetic transaminase (SGOT), alkaline phosphatase, and total bilirubin. Each laboratory value will be categorized as follows:

- < 1.5 × ULN
- $\geq 1.5 \times ULN < 3.0 \times ULN$



- $\geq 3.0 \times ULN < 5.0 \times ULN$
- $\geq 5.0 \times \text{ULN} < 10.0 \times \text{ULN}$
- $\geq 10.0 \times \text{ULN} < 20.0 \times \text{ULN}$
- $\geq 20.0 \times ULN$

Shift tables of Baseline to the maximum (relative to the normal range, i.e., the largest multiple relative to the upper limit of normal) values, and from Baseline to final value will be presented using these categories. A listing of potentially clinically important liver function laboratory values will be provided. The listing will include all subjects who met any of the following four criteria:

- ALT  $\geq$  3 × ULN, or
- AST  $\geq$  3 × ULN, or
- Alkaline phosphatase  $\geq 1.5 \times ULN$ , or
- Total bilirubin  $\geq 2 \times ULN$ .

A listing of possible Hy's Law cases, defined as those who meet all of the following conditions will be provided:

- ALT  $> 3 \times ULN$  or AST  $> 3 \times ULN$
- Associated with an increase in bilirubin  $\geq 2 \times ULN$
- Alkaline phosphatase  $< 2 \times ULN$ .

#### 11.4 Analysis of Vital Signs and Weight

## 11.4.1 Variables and Criteria Defining Abnormality

The following vital sign parameters will be assessed: Systolic blood pressure [mmHg], Diastolic blood pressure [mmHg], Pulse [beats per minute], Respiratory rate [breaths per minute], Temperature [°C], Weight [kg]. The following table presents the Criteria for Potentially Clinically Important Vital Sign Findings. Of note, a post baseline value must



be more extreme than the baseline value to be considered a potentially clinically important finding.

Table 15. Criteria for Potentially Clinically Important Vital Sign Findings

| Vital Sign | Category | Criteria for Potential Clinically Important Vital Signs |
|---|---|---|
| Systolic Blood Pressure | Low Value | $\leq 90$ mmHg and decrease $\geq 20$ mmHg from Baseline |
| | High Value | $\geq 160 \mbox{ mmHg}$ and increase $\geq 20 \mbox{ mmHg}$ from Baseline |
| Diastolic Blood Pressure | Low Value | ≤ 50 mmHg and decrease ≥ 15 mmHg from Baseline |
| | High Value | $\geq 105$ mmHg and increase $\geq 15$ mmHg from Baseline |
| Pulse Low Value | | ≤ 50 bpm and decrease ≥ 15 bpm from Baseline |
| | High Value | ≥ 120 bpm and increase ≥ 15 bpm from Baseline |

#### 11.4.2 Statistical Methods

Changes from Baseline to each visit and to the final value in vital sign parameters will be summarized with the mean, standard deviation and median. The Baseline and final value means will also be presented for subjects who have both the Baseline and final values (see Section 6.0 for the definition of Baseline and final values).

For baseline, if there are multiple measurements on the same day, the last measurement prior to the first dose of study drug will be used as the Baseline vital sign value. If there are multiple post-baseline measurements on the same day, average value will be used.

For systolic blood pressure, diastolic blood pressure and pulse, a listing of all subjects with any vital sign value meeting criteria for potentially clinically important values will be provided. For each of these subjects, the whole course of the respective parameter will be listed. The number and percentage of subjects who have at least one value meeting criteria for potentially clinically important values will be provided for each selected vital sign parameter.

All analyses will be conducted in the Safety Population. Table for potentially clinically important vital signs will also be summarized in the ALL RZB Population.



#### 11.5 Analysis of ECG Parameters

The ECG parameters will be assessed as scheduled in the study protocol.

Summary statistics for mean change from baseline for corrected QT interval (QTc) using Bazett (QTcB) and Fridericia (QTcF) corrections, aggregated, will be provided by analysis visits.

- Values for both QTcF and QTcB interval measurements will be categorized into the following: ≤ 450 ms, > 450 ms, > 480 ms, > 500 ms, or missing. For the scheduled visits, as well as baseline, the number and percentage of subjects within each category will be presented. Additionally, for each category, the number and percentage of subjects with a maximum QTcF interval falling into the category will be presented; a similar summary will be presented for QTcB intervals.
- For QTcF and QTcB intervals, the changes from baseline will be categorized into the following: < 30 ms, 30 ≤ − < 60 ms, ≥ 60 or missing. For the scheduled visits, the number and percentage of subjects within each category will be presented. Additionally, for each category, the number and percentage of subjects with a maximum change from baseline in the QTcF interval falling into the category will be presented; a similar summary will be presented for QTcB intervals.

Analyses will be conducted in the Safety Population.

#### 11.6 Local Tolerability

Local tolerability at the administration site of the subcutaneous injection will be assessed by the investigator in the measurements of "swelling," "induration," "heat," "redness," "pain," or "other findings."

Proportion of subjects reporting each condition will be analyzed. The overall rate (with at least one occurrence) during Part A and B will also be presented.

Analyses will be conducted in the Safety Population in Part A and in Part B.

## 12.0 Pharmacokinetic Analysis

Pharmacokinetic analysis is not covered in this SAP.

## 13.0 Biomarkers Analysis

Biomarkers Analysis is not covered in this SAP.

| 14.0 | Summary of Changes |
|---|---|
| 14.1 | Summary of Changes Between the Latest Version of Protocol and the Current SAP |

14.2 Summary of Changes Between the Previous Version and the Current Version of the SAP

15.0 Appendix

None.

16.0 References

None.

17.0 List of Tables, Figures, and Data Listings to Be Programmed

To be provided in a separate document.

## **Document Approval**

Study M16004 - Statistical Analysis Plan Version 1 - 10Jan2018 (E3 16.1.9)

Version: 2.0 Date: 10-Jan-2018 11:00:31 PM Company ID: 01102018-00F9F683BCCDCD-00002-e

| Signed by: | Date: | Meaning Of Signature: |
|------------|-------------------------|-----------------------|
| | 10-Jan-2018 05:32:25 PM | Author |
| | 10-Jan-2018 06:24:16 PM | Approver |
| | 10-Jan-2018 07:10:00 PM | Approver |
| | 10-Jan-2018 11:00:30 PM | Approver |